CLINICAL TRIAL: NCT07390435
Title: Feasibility and Acceptability of Collecting Sociodemographic Data in CCTG Trials
Status: Not yet recruiting | Type: Observational
Sponsor: Canadian Cancer Trials Group (Network)
Responsible Party: Sponsor
Other Study IDs: SC32S
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Social Determinants of Health Questionnaire — This study will use a standardized SDoH Questionnaire to collect the required sociodemographic data

SUMMARY:
This study is being done to answer the following question: Are patients on a clinical trial willing to provide answers to questions about their social, economic, and environmental factors-sometimes called social determinants of health-which affect people's health experiences and access to care. These factors may include income, education, employment, housing, social supports, and experiences with discrimination or stress. Participation will help researchers better understand barriers to participating in clinical trials and access to health care.

DETAILED DESCRIPTION:
It is anticipated that 1000 people will take part in this study. Participation in this study will only take about 10 minutes or less. Participants who choose to take part in this study will be asked to fill out a form with questions in English or French about the non-medical factors that influence health. This includes asking about the conditions and places in which the participant lives, learns, works, and plays. Participants will also be asked how they feel about answering these questions. Researchers will use this information to better understand who participates in clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) with cancer who are either:

  * Currently being screened and consented to a CCTG trial (prospective).
  * Already enrolled in an ongoing CCTG trial and still under follow-up (retrospective).

Exclusion Criteria:

* Participants already enrolled or expected to enroll in a CCTG trial that is also collecting the SDoH Questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is designed to include participants who have consented to a CCTG clinical trial. If a patient consents to a CCTG trial but does not enroll, they will remain eligible for SC.32S.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the feasibility of collecting comprehensive sociodemographic data via a standardized SDoH Questionnaire among participants being screened and consented to a CCTG trial and participants already enrolled in a CCTG trial | 12 months

SECONDARY OUTCOMES:
To assess the acceptability of this SDoH questionnaire to participants. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Leah Lambert, Study Chair — BCCA - Vancouver Cancer Centre, Vancouver, BC Canada; Michael McKenzie, Study Chair — BCCA - Vancouver Cancer Centre

IPD SHARING:
Plan to Share IPD: Yes
As per CCTG policy.
URL: https://www.ctg.queensu.ca/public/policies